CLINICAL TRIAL: NCT06664294
Title: The USE of ULTRASONOGRAPHY in CONFIRMING SUPRAGLOTTIC AIRWAY DEVICE PLACEMENT in PEDIATRIC PATIENTS
Status: Active, not recruiting | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Busra Yaka, principal investigator, Kocaeli University
Other Study IDs: KAEK2024/171
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Airway Ultrasound
Keywords: supraglottic airway pediatric airway,airway ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In this study,the investigators evaluated the placement of the supraglottic airway device with ultrasonographic imaging.

DETAILED DESCRIPTION:
After informing the patients about the study and possible risks, written consent was obtained from all patients. After routine anesthesia technique was applied to the patients, supraglottic airway device was inserted. The placement of the airway device was evaluated with ultrasonography. Airway pressures reflected on the anesthesia device were recorded. The correlation between airway pressures and ultrasonographic images was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with informed consent from their parents
* Patients with ASA I-II physical status
* Patients with appropriate fasting time
* Those with an operation time of less than 2 hours

Exclusion Criteria:

* ASA III-IV physical status patients
* Patients with respiratory tract infections
* Patients undergoing head and neck surgery
* Patients with oropharyngeal pathology
* Patients with gastrointestinal obstruction
* Patients with tracheomalacia
* Patients who need to be intubated for anesthesia applications

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric patients aged 3-15 years with an operation time of less than 2 hours
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2025-01-29 (Estimated); Study Completion 2025-04-29 (Estimated)

PRIMARY OUTCOMES:
correlation between ultrasonography and clinical tests | 24 hours
  Our primary aim was investigation of correlation between ultrasonography and clinical tests for placement of supraglottic airway device in pediatric patients.

SECONDARY OUTCOMES:
mesuring airway pressures | 24 hours
  Our secondary aim was measuring airway pressures, measuring the difference between the tidal volume delivered from the anesthesia device and the volume withdrawn from the patient, and its correlation with correct placement

CONTACTS AND LOCATIONS:
Overall Officials: can aksu, Study Director — Kocaeli University
Locations (1):
- Kocaeli University, İzmit, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Çalışmanın kopyalanmasının önüne geçmek için

REFERENCES:
- [Background] Kim J, Kim JY, Kim WO, Kil HK. An ultrasound evaluation of laryngeal mask airway position in pediatric patients: an observational study. Anesth Analg. 2015 Feb;120(2):427-32. doi: 10.1213/ANE.0000000000000551. PMID 25545750